CLINICAL TRIAL: NCT01494259
Title: Use of Percutaneously-Placed Continuous Flow Bupivacaine Pain Pumps to Decrease Post-operative Pain Following Mastectomy With Immediate Reconstruction: A Prospective, Randomized, Double-Blind Clinical Trial
Brief Title: Bupivacaine Pain Pumps to Decrease Mastectomy Post-Operative Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Gedge Rosson, Associate Professor, Dept. of Plastic and Reconstructive Surgery; Director of Breast Reconstruction, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00010363
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: immediate breast reconstruction; pain control; post mastectomy pain control
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine; Epinephrine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Treatment) Group (Experimental): The Symbios GOPump is the Food and Drug Administration-approved delivery device used to infuse the bupivacaine. The pump is attached to catheters placed in the patient's breast reconstruction site. A 10cm long 16-guage needle is provided to aid insertion of the catheter into the patient. The entire catheter will pass through the bore of the introducer needle. A 60cc syringe is used to fill the Symbios GOPump through the fill port. After filling the 60cc syringe with up to 300cc of 0.5% bupivacaine, the syringe is attached to the port and the medication injected into the infusion pump. The steady-flow pressure regulator maintains a constant 6 psi pressure in the outflow chamber ensuring a uniform flow of medication through each catheter inserted into the Symbios GOPump.
  Interventions: Drug: Bupivacaine
- Saline (Placebo) Group (Placebo Comparator): The Symbios GOPump is the Food and Drug Administration-approved delivery device used to infuse the saline. The pump is attached to catheters placed in the patient's breast reconstruction site. A 10cm long 16-guage needle is provided to aid insertion of the catheter into the patient. The entire catheter will pass through the bore of the introducer needle. A 60cc syringe is used to fill the Symbios GOPump through the fill port. After filling the 60cc syringe with up to 300cc of normal saline, the syringe is attached to the port and the medication injected into the infusion pump. The steady-flow pressure regulator maintains a constant 6 psi pressure in the outflow chamber ensuring a uniform flow of medication through each catheter inserted into the Symbios GOPump.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — Up to 300cc of 0.5% bupivacaine administered to the mastectomy site via 2 catheters connected to the Symbios GOPump at a rate of 2 cc per hour per catheter over 3 days.
  Other Names: Marcaine with epinephrine
  Arms: Bupivacaine (Treatment) Group
Drug: Saline — Up to 300cc of normal saline administered to the mastectomy site via 2 catheters connected to the Symbios GOPump at a rate of 2 cc per hour per catheter over 3 days.
  Other Names: Normal Saline
  Arms: Saline (Placebo) Group

SUMMARY:
This double-blind, randomized, controlled clinical trial comparing patient-reported pain and pain medication/narcotic use between patients randomized to treatment (bupivacaine) or placebo (saline) delivered via pain pump to the mastectomy site. Candidates will have chosen to have a mastectomy on one side immediately followed with tissue expander placement breast reconstruction.

Patients will be randomized 1:1 to bupivacaine- (treatment) or saline-(placebo) filled percutaneously-placed pain pumps; neither the participants nor the study staff will know participants' treatment. Data on patient-perceived pain and pain medication use will be collected before surgery, during surgery, and after surgery on Days 1, 2, 3, 7, and 90, and at Years 2 and 4 by phone.

The investigators hypothesize that patients randomized to the treatment (bupivacaine) group will have significantly lower pain scores and use less pain medicine than patients who receive placebo during the first 90 days following their surgery. The Year 2 and Year 4 follow-ups are included as tertiary endpoints to capture differences in chronic pain, and patients will be asked to complete the same questionnaires as at the Day 90 follow up.

DETAILED DESCRIPTION:
Double-blind, randomized, controlled clinical trial comparing patient-reported pain and pain medication/narcotic use between patients randomized to treatment (bupivacaine) or placebo (saline) delivered via pain pump to the mastectomy site. Candidates will have elected to undergo unilateral post-mastectomy immediate tissue expander breast reconstruction. Participants meeting inclusion criteria will be enrolled and baseline data collection completed prior to randomization and surgery.

Patients will be randomized 1:1 to bupivacaine- (treatment) or saline-(placebo) filled percutaneously-placed pain pumps in a double-blinded design. Patient-specific surgical details will be recorded intraoperatively. Following the surgery, post-operative pain, pain medication/narcotic use, and assessment for adverse events (AEs)/serious adverse events (SAEs) will be assessed on Days 1, 2, and 3. A clinic visit occurs on Day 7 when the pain pump will be removed and additional data collected (updated medical history, pain medication/narcotic use, AEs/SAEs, and study questionnaires). A Pain Pump Questionnaire will be completed to obtain the patient's assessment of the usability of the pain pump.

Long-term quality-of-life/health outcomes assessments will be done on post-operative Day 90 (±14 days), Year 2 (±14 days), and Year 4 (±14 days). The Year 2 and Year 4 follow-ups are included as tertiary endpoints to capture differences in chronic pain, and patients will be asked to complete the same questionnaires as at the Day 90 follow up.

ELIGIBILITY:
Inclusion Criteria:

* Be Female aged 18-100 years.
* Choose unilateral mastectomy followed by immediate tissue expander breast reconstruction.
* Have no inflammatory breast cancers.
* Be aware of the nature of her malignancy.
* Understand the study purpose, requirements, and risks.
* Be able and willing to give informed consent.

Exclusion Criteria:

* Any concurrent narcotic analgesic use (baseline narcotic use must be 0 to be eligible).
* Axillary lymph node dissection related to qualifying mastectomy.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Differences in post-operative static and moving pain scores between patients randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control. | Day of Surgery through Day 7
  Post-operative pain, pain medication/narcotic use, and assessment for adverse events (AEs)/serious adverse events (SAEs) will be assessed the Day of surgery through post-operative Day 7. A clinic visit occurs on Day 7 when the pain pump will be removed and additional data collected (updated medical history, pain medication/narcotic use, AEs/SAEs, and study questionnaires).

SECONDARY OUTCOMES:
Document long-term changes in QOL scores between patients randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control. | Day 90
  Document long-term changes in Quality of Life (QOL) scores [the RAND-36 Health Survey, Disability of the Arm, Shoulder, and Hand (Quick DASH) questionnaire, and Breast-Q scores] between women undergoing unilateral mastectomy followed by unilateral immediate tissue expander breast reconstruction randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control.
Document long-term changes in QOL scores between patients randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control. | Year 2
  Document long-term changes in Quality of Life (QOL) scores [the RAND-36 Health Survey, Disability of the Arm, Shoulder, and Hand (Quick DASH) questionnaire, and Breast-Q scores] between women undergoing unilateral mastectomy followed by unilateral immediate tissue expander breast reconstruction randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control.
Document long-term changes in QOL scores between patients randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control. | Year 4
  Document long-term changes in Quality of Life (QOL) scores [the RAND-36 Health Survey, Disability of the Arm, Shoulder, and Hand (Quick DASH) questionnaire, and Breast-Q scores] between women undergoing unilateral mastectomy followed by unilateral immediate tissue expander breast reconstruction randomized either to bupivacaine- (treatment) or saline- (placebo) filled, percutaneously-placed pain pump analgesic administration for post-operative pain control.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Plastic and Reconstructive Surgery, Johns Hopkins, Baltimore, Maryland, United States